CLINICAL TRIAL: NCT01487317
Title: A Randomized, Double-blind, Placebo-controlled Study of an Acetylcholinesterase Inhibitor in the Management of Delirium in Hospitalized Patients Aged 75 Years and Over
Brief Title: Rivastigmine in the Management of Delirium
Acronym: confuriv
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P071244; 2009-015632-15 (EudraCT Number)
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Delirium
Keywords: Delirium; acetylcholinesterase inhibitor; Elderly; Emergency department
MeSH Terms: conditions — Delirium; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivastigmine transdermal patch (Experimental)
  Interventions: Drug: Rivastigmine transdermal patch
- placebo (Placebo Comparator)
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: Rivastigmine transdermal patch — One transdermal patch of Rivastigmine (equivalent to 4.6 mg/24h per os) per day from randomization to day 14 before day 14: end od treatment, if DRS R-98 severity < 10 during 2 consecutive days At day 14, if DRS R-98 severity ≥ 10: one transdermal patch of Rivastigmine 9.5 mg/24h per day from day 14 to day 30 if DRS R-98 severity < 10, the active treatment will be stopped
  Arms: Rivastigmine transdermal patch
Drug: placebo patch — One transdermal patch of placebo per day from randomization to day 14 Before day 14: end of treatment if DRS R-98 severity < 10 during 2 consecutive days, At day 14 if DRS R-98 severity ≥ 10: One transdermal patch of placebo per day from day 14 to day 30 if DRS R-98 severity < 10, the placebo treatment will be stopped
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the efficacy of an anticholinesterase treatment in patients aged 75 and over, hospitalized with delirium.

Study type : Interventional Study design: randomized, double-blind, placebo-controlled study during one month and a 11-month follow-up

DETAILED DESCRIPTION:
Delirium affects up to 50% of hospitalized patients aged 75 and over. Delirium increases risk of comorbid illness, hospital length of stay, institutionalization, and death. Patients with diagnosed or undiagnosed cognitive impairment are at risk to develop delirium. In a prospective study, half of elderly patients with delirium seen in the emergency department had cognitive impairment.

Hypothesis: cholinesterase inhibitors reduce duration and severity of delirium

Main objective:

- to assess the efficacy of cholinesterase inhibitors in patients aged 75 and over hospitalized with delirium

Secondary objectives:

* to describe at one year the percentage of these patients who have a diagnosis of Alzheimer's disease and associated disorders
* to assess the sensitivity to cholinesterase inhibitors in the sub-group of patients with a diagnosis of dementia at one year Design and methods Multicenter, randomized, controlled study with two parallel arms: a rivastigmine group and a placebo group. The study includes a treatment period of one month and a follow-up of 11 months.

Evaluation of the delirium severity will be conducted with DRS-R98 severity each day during the hospitalization.

At day 14, according to DRS-R98 severity score, interruption of treatment or upward dose titration At day 30, last treatment (active or placebo) administration and evaluation with CAM, DRS-R98 severity, MMSE and DSM IV dementia criteria. In case of dementia diagnosis, investigator (MD) will identify the etiologic diagnosis.

At month 3 and 12, evaluation with CAM, DRS-R98 severity, MMSE and DSM IV dementia criteria, number of consultation and hospitalization. In case of dementia diagnosis, , investigator (MD) will identify the etiologic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 and over
* Hospitalization for delirium not correlated to surgery for less than 48 hours
* Patients with delirium requiring the presence of features 1 (acute onset and fluctuation course), 2 (inattention), 3 (disorganized thinking) and 4 (altered level of consciousness) of the Confusion Assessment Model and DRS R-98 > 10
* Absence of any contraindications to a cholinesterase inhibitor treatment
* Health insurance affiliation
* Having signed an informed consent form
* Caregiver/informant to provide information on patient

Exclusion Criteria:

* Use of IAchE or memantine medication
* Contraindication to IAchE medication
* Frontotemporal dementia
* Diseases involving the short-term survival
* Digestive bleeding
* Ischemic and hemorrhagic stroke related to actual onset (including hemorrhagic contusion)
* Natremia ≤120 mmol/l at the time of hospitalization
* Post epileptic confusion
* Hepato-cellular failure
* Cardiorespiratory impairment at risk of transfer to intensive care unit
* Major sensory deficits that could interfere with cognitive assessment (visual and auditory)
* Not fluent in French
* Being under guardianship
* Absence of caregiver/informant to sign informed consent form

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay from randomization to declaration by investigator (MD) that patient can leave acute care | to a maximum of 12 months

SECONDARY OUTCOMES:
Percentage of patients with persistent delirium symptoms (DRS R-98 scale) | at day 14
Percentage of patients with persistent delirium symptoms (DRS R-98 scale) | at day 30
Percentage of patients with persistent delirium symptoms at day 30 (CAM scale) | at day 30
Percentage of patients with a dementia diagnosis at 12 months (according to the DSM IV criteria) | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Verny, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié Salpetriere Hospital, Paris, France